CLINICAL TRIAL: NCT06856915
Title: Effects of Home-based Respiratory Muscle Training by Telerehabilitation on Quality of Life, Cardiopulmonary Function, Physical Status and Psychological Status in Individuals With Ischemic Heart Disease
Brief Title: Effects of Home-based Respiratory Muscle Training Progamme in Individuals With Ischemic Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Instituto de Investigación Sanitaria Hospital Clínico San Carlos (Unknown); European Regional Development Fund (Other); Hospital Universitario 12 de Octubre (Other)
Responsible Party: Principal Investigator, Ibai López de Uralde Villanueva, Tenure-track professor with a PhD in the Department of Radiology, Physiotherapy and Rehabilitation, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PI23/00816
Record Dates: First submitted 2025-01-20; First posted 2025-03-04 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Ischemic Heart Disease
Keywords: Respiratory muscle training; Cardiac rehabilitation; Quality of Life; cardiopulmonary function; physical state; psychological state; Telerehabilitation
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Inspiratory muscle training group + Exercise training (Active Comparator): Participants in this group will perform a home-based inspiratory muscle training programme (8 weeks) by telerehabilitation and after a center-based conventional cardiovascular exercise programme (8 weeks)
  Interventions: Other: Inspiratory muscle training; Other: Conventional cardiac rehabilitation programme
- Inspiratory muscle training sham group + Exercise training (Sham Comparator): Participants in this group will perform a home-based sham inspiratory muscle training programme (8 weeks) by telerehabilitation and after a center-based conventional cardiovascular exercise programme (8 weeks)
  Interventions: Other: Sham inspiratory muscle training; Other: Conventional cardiac rehabilitation programme
- Inspiratory and expiratory muscle training group + Exercise training (Experimental): Participants in this group will perform a home-based inspiratory and expiratory muscle training programme (8 weeks) by telerehabilitation and after a center-based conventional cardiovascular exercise programme (8 weeks)
  Interventions: Other: Combined inspiratory and expiratory muscle training; Other: Conventional cardiac rehabilitation programme
- Inspiratory and expiratory muscle training Sham group + Exercise training (Sham Comparator): Participants in this group will perform a home-based sham inspiratory and expiratory muscle training programme (8 weeks) by telerehabilitation and after a center-based conventional cardiovascular exercise programme (8 weeks)
  Interventions: Other: Sham combined inspiratory and expiratory muscle training; Other: Conventional cardiac rehabilitation programme

INTERVENTIONS:
Other: Inspiratory muscle training — Participants will engage in inspiratory muscle training programme at home using an inspiratory muscle training threshold device . This training will be conducted twice daily, five days a week, for eight weeks, with physiotherapist supervision provided three times per week by telerehabilitation.
  Arms: Inspiratory muscle training group + Exercise training
Other: Combined inspiratory and expiratory muscle training — Participants will engage in inspiratory+expiratory muscle training programme at home using an inspiratory+expiratory muscle training threshold device . This training will be conducted twice daily, five days a week, for eight weeks, with physiotherapist supervision provided three times per week by telerehabilitation.
  Arms: Inspiratory and expiratory muscle training group + Exercise training
Other: Sham inspiratory muscle training — Participants will engage in sham inspiratory muscle training programme at home using a sham inspiratory muscle training threshold device . This training will be conducted twice daily, five days a week, for eight weeks, with physiotherapist supervision provided three times per week by telerehabilitation.
  Arms: Inspiratory muscle training sham group + Exercise training
Other: Sham combined inspiratory and expiratory muscle training — Participants will engage in sham inspiratory+expiratory muscle training programme at home using a sham inspiratory+expiratory muscle training threshold device . This training will be conducted twice daily, five days a week, for eight weeks, with physiotherapist supervision provided three times per week by telerehabilitation.
  Arms: Inspiratory and expiratory muscle training Sham group + Exercise training
Other: Conventional cardiac rehabilitation programme — Following the respiratory muscle training programme, participants will transition to a center-based cardiovascular exercise programme conducted twice weekly for eight weeks.

SUMMARY:
The main objective of the present study is to verify whether respiratory muscle training programme (IMT+EMT; included both inspriratory and expiratory muscles), applied by telerehabilitation, is an effective intervention (versus placebo and versus inspiratory muscle training in isolation (IMT)) in improving quality of life, cardiopulmonary function and physical and psychological state in people with ischemic heart disease. In addition, the aim is to determine whether respiratory muscle training (IMT or IMT+EMT) is effective in enhancing the results obtained by a conventional cardiac rehabilitation programme on the aforementioned variables.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ischemic heart disease
* Age 18 years or older
* Cardiovascular clinical stability

Exclusion Criteria:

* Any condition that contraindicate exercise training
* Inability to close the lips to hold the training device's mouthpiece (e.g., facial paralysis)
* Previous participation in a rehabilitation programme within the last 3 months
* Pregnancy
* Inability to adhere to remote monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  EuroQol-five-dimensional Questionnaire A numerical value represented Health state as EQ-5D 'index values' or 'index scores' reflecting how good or bad a health state is.
  The VAS is a scale from 0 (worst imaginable health state) to 100 (best imaginable health state).

SECONDARY OUTCOMES:
Modified Medical Research Council Dyspnoea Scale | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  The modified Medical Research Council (mMRC) assess the degree of functional disability due to dyspnoea. The mMRC breathlessness scale ranges from grade 0 to 4. Higher scores mean a worse dyspnoea.
Fatigue | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  Multidimensional Fatigue Inventory (MFI-17) The MFI is a valid and reliable instrument for assessing fatigue severity. It consists in 17 items ranked from 1 to 5, the maximun value is 85 points and the minimum 17 points. Higher scores mean a worse fatigue.
Cardiopulmonary function: level of exercise capacity | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  Exercise capacity will be measured using a Cardiopulmonary exercise testing (CPET) that precisely defines maximum exercise capacity through measurement of peak oxygen uptake. The following parameters will be acquired by breath-by-breath analysis using an automated gas analyzer: minute ventilation rate; oxygen consumption (VO2); carbon dioxide production (VCO2); and the other variables of to assess aerobic capacity and to identify potential limiting factors.
  An electrocardiogram and blood pressures will be recorded at rest, throughout exercise and during recovery.
Strength and endurance of the lower limbs | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  1 minute sit to stand
Upper limb strenght | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  Upper limb muscle strength (handgrip force) will be assessed using a hand-held dynamometer. Three measurements will be performed for each hand, alternating sides, with the elbow at 90° flexion. The best value will be recorded in kilogrames.
Respiratory muscle strength | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  Maximal inspiratory preassure and Maximal expiratory preassure
Inspiratory muscle endurance | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  Inspiratory muscle endurance will be assed by an incremental load test that required subjects to breathe against inspiratory threshold loads that were increased each minute by 10% of baseline PI,max until voluntary task failure muscle endurance test. Inspiratory muscle endurance was defined as the PI,max sustained for a minimum of 1 min.
Anxiety and depression levels | Pre -intervention, at the end of the respiratory muscle training (8 weeks) and post intervention(16 weeks)
  The Hospital Anxiety and Depression Scale (HADS) is a self-assessment questionnaire for detecting states of anxiety and depression. The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level.

CONTACTS AND LOCATIONS:
Locations (1):
- Departamento de Radiología, Rehabilitación y Fisioterapia, Facultad de Enfermería, Fisioterapia y Podología, Universidad Complutense de Madrid, Madrid, Madrid, Spain